CLINICAL TRIAL: NCT06338254
Title: Efficacy of Percussion Massage Therapy Applied to the Lower Extremity on Pain, Edema, and Quality of Life in Pregnant Women: Randomized Controlled Trial
Brief Title: Efficacy of Percussion Massage Therapy Applied to the Lower Extremity on Pain, Edema in Pregnant Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, merve yilmaz menek, Principal Investigator, Istanbul Medipol University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: E-10840098-772.02-5416
Record Dates: First submitted 2024-03-14; First posted 2024-03-29 (Actual); Last update posted 2024-03-29 (Actual); Status verified 2024-03

CONDITIONS: Pregnancy Complications; Edema Leg; Physiotherapy
Keywords: Edema; pain; percussion massage therapy; pregnancy; quality of life
MeSH Terms: conditions — Pregnancy Complications; Edema; Pain

STUDY DESIGN:
Who Masked: Participant
Masking Description: The participants are blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PMT Group (Experimental): Pregnant women included in this group received a total of 12 sessions of percussion massage therapy, applied to their bilateral lower extremities for four weeks.
  Interventions: Other: percussion massage therapy
- Control Group (No Intervention): No massage therapy was applied to the lower extremities of the pregnant women in this group.

INTERVENTIONS:
Other: percussion massage therapy — Pregnant women included in this group received a total of 12 sessions of percussion massage therapy, applied to their bilateral lower extremities for four weeks. Percussion massage was applied to both extremities at separate times for 5 minutes each with the Hypervolt device. (Fig. 2) Four muscles in total were focused on; These muscles are medial gastrocnemius, lateral gastrocnemius, peronus longus, and tibialis anterior. Percussion massage was applied in the longitudinal direction of the muscle, from distal to proximal and back to distal, going from posterior to anterior muscle groups. Percussion massage started on the medial side and ended on the lateral side for each muscle. Equal pressure and duration were applied to each muscle.
  Arms: PMT Group

SUMMARY:
This study aim is to examine the effect of percussion massage therapy applied to lower extremity on pain, edema, fatigue and quality of life in pregnant women.

DETAILED DESCRIPTION:
Aim: This study aim is to examine the effect of percussion massage therapy applied to lower extremity on pain, edema, fatigue and quality of life in pregnant women.

Methods: Sixty pregnant women between 24 and 36 weeks of pregnancy were included in the study. Pregnant women were randomly divided into two groups: The percussion massage treatment (PMT) group and the control group. Pregnant women included in the PMT group received a total of 10 sessions of percussion massage therapy, applied to their bilateral medial gastrocnemius, lateral gastrocnemius, peronus longus and tibialis anterior muscles three times a week. No massage therapy was applied to the lower extremities of the pregnant women in the control group. Pain assessment with Visual analog scale (VAS), ankle, knee, and thigh circumference measurements with tape measure, fatigue level with Fatigue Severity Scale (FSS), and quality of life assessment with Short Form- 36 (SF-36) were conducted.

ELIGIBILITY:
Inclusion Criteria:

* being pregnant between the ages of 18-40,
* being in the 24-36 weeks of pregnancy,
* not being at risk of pregnancy,
* being pregnant with a single baby,
* having complaints of pain or edema in the lower extremities,
* volunteering to participate in the study 3 days a week

Exclusion Criteria:

* multiple pregnancies,
* pregnant women with anemia,
* presence of circulatory problems,
* cardiovascular disease,
* chronic orthopedic disease,
* foot-related orthopedic and vascular disease.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2022-09-04 (Actual); Primary Completion 2023-06-04 (Actual); Study Completion 2023-06-10 (Actual)

PRIMARY OUTCOMES:
The Visual Analog Scale (VAS) | 5 minutes
  The VAS is a single-item scale with a line length of 10 cm. In this line, 0 means "I have no pain," whereas 10 means "worst pain" at the end. Participants were asked to indicate on a 10-point scale how much discomfort they were experiencing
Evaluation of edema | 10 minutes
  Measurement was made with a non-flexible tape measure. Care was taken not to compress the tissues during measurement. The patient should be in a comfortable position on his back. The measurement was made with a tape measure, on the medial and lateral malleolar areas for the foot, on the midline of the patella for the knee, and the widest area for the calf and thigh.
Fatigue Severity Scale (FSS) | 5 minutes
  It includes the evaluation of the severity and timing of fatigue and the effects of fatigue on daily activities in individuals. It covers the fatigue severity of individuals in the last month. Each question on the scale is scored between 1 and 7 and contains nine questions in total. The arithmetic average of all scores was taken
Short Form-36 (SF-36) | 15 minutes
  The test that consists of 36 items and evaluates 8 subheadings assess the level of quality of life. It includes testing of physical and social function, role limitations due to physical and emotional problems, pain, mental health, energy, and finally general perception of health. The second question of the scale covers the 12-month evaluation and the remaining questions cover the last month. The questions are Likert-type, except for the fourth and fifth questions. The score is calculated by reversing items 1, 6, 7, 8, 9a, 9d, 9e, 9h, 11b, 11d of the scale. The score covers the range from 0 to 100. While 0 describes poor health, 100 describes good health

CONTACTS AND LOCATIONS:
Overall Officials: MERVE YILMAZ MENEK, PhD, Principal Investigator — Medipol University
Locations (1):
- Istanbul Medipol University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
It is not to planned to share individual participant data (IPD)

REFERENCES:
- [Result] Coban A, Sirin A. Effect of foot massage to decrease physiological lower leg oedema in late pregnancy: a randomized controlled trial in Turkey. Int J Nurs Pract. 2010 Oct;16(5):454-60. doi: 10.1111/j.1440-172X.2010.01869.x. PMID 20854342
- See also: Effect of foot massage to decrease physiological lower leg oedema in late pregnancy: a randomized controlled trial in Turkey — https://pubmed.ncbi.nlm.nih.gov/20854342/